CLINICAL TRIAL: NCT04330378
Title: A Hospital-at-Home Pilot in Singapore: A Prospective Quasi-Experimental Cohort Study
Brief Title: A Hospital-at-Home Pilot in Singapore
Status: Completed | Type: Observational
Sponsor: National University Health System, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Stephanie Ko, Associate Consultant, National University Health System, Singapore
Other Study IDs: 2020/00345
Record Dates: First submitted 2020-03-27; First posted 2020-04-01 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Hospital-at-home
Keywords: Home Care; Hospital-in-the-home; Home Hospital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hospital-at-home: All patients who are enrolled into the NUHS@Home Programme will be recruited into this arm. Patients will be sent home via ambulance, where they will be reviewed by a NUHS@Home nurse. Intravenous therapies, pillboxes for medication, remote monitoring software, and telecommunication tools will be set up as indicated. NUHS@Home doctors will visit at least once daily, and nurses at least twice daily as required. Therapists will conduct home visits as necessary. The NUHS@Home team is available 24/7. When conventional discharge criteria are met, the patient will be discharged. The NUHS@Home clinical team will be under clinical governance of Division of Advanced Internal Medicine at NUH and patients will be considered 'inpatients' throughout the treatment period.
  Interventions: Other: Hospital-at-home
- Usual in-hospital care: Patients who would otherwise be eligible for NUHS@Home but are not able to be enrolled due to capacity will be recruited into this arm. They will receive usual care in the wards that they are already in until they are discharged.
  Interventions: Other: Usual in-hospital care
- Rejected cohort: Patients who were offered but declined enrolments inot the NUHS@Home programme will be approached for consent to be in the rejected cohort. There will be no change to the patient's clinical management.
  Interventions: Other: Usual in-hospital care

INTERVENTIONS:
Other: Hospital-at-home — As per experimental arm
  Other Names: Home Hospitalisation; Home Hospital; Hospital-in-the-home
  Groups: Hospital-at-home
Other: Usual in-hospital care — As per control arm
  Groups: Rejected cohort; Usual in-hospital care

SUMMARY:
Hospital-at-home models seek to address the impending shortage of hospital beds by reimagining the way we deliver acute hospital-level care - substituting the ward for a patient's home. Such programmes have been well established in other countries such as Australia, Europe and USA to be a less costly way to provide inpatient care as a result of a reduction of fixed costs of building and running hospitals, with equivalent variable costs and comparable clinical outcomes. Acute services are provided at home, including regular visits by doctors, nurses and therapists, intravenous therapy, simple investigations and 24/7 access to doctors. The clinical service is tech-enabled, by remote monitoring and telecommunication technologies.

Although overseas experience suggests that hospital-at-home programmes are an effective, safe and scalable substitute for inpatient beds, and promising strategy to meet the bed demands of our ageing population, the outcomes in the local environment is unclear. Singapore has a unique healthcare system compared to primarily insurance driven (USA) or publicly funded (UK and Australia), which favours subsidies of inpatient care compared to community-based care. In addition, cultural beliefs of hospitals as a source of comfort and healing and unfamiliarity with healthcare providers performing home visits may provide unique challenges which may affect outcomes of a hospital-at-home programme in Singapore. In an Asian setting, family and informal caregivers are heavily involved in the care of patients and may pose unique barriers and facilitators to such care at home that may not be evident in similar models in Western countries.

This study aims to evaluate the effectiveness, feasibility and processes of a new hospital-at-home programme in Singapore.

DETAILED DESCRIPTION:
1. Hypothesis

   We hypothesise that hospital-at-home programmes may reduce cost of delivering care with comparable clinical outcomes (readmissions, mortality, and hospital-acquired complications) and positive patient and staff experiences.
2. Specific Aims

The primary objective of this study is:

1. To compare the mean direct cost of care per day of index hospitalisation for patients receiving HaH care to similar patients receiving usual inpatient care.

The secondary objectives in this study are:

1. To evaluate the clinical effectiveness, in terms of 30-day readmissions, mortality and hospital-acquired complications) of HaH compared to usual inpatient care;
2. To evaluate impact of patient-reported outcomes (EQ-5D, Care Transitions Measure and patient satisfaction scores) of HaH compared to usual inpatient care, including impact on medication management;
3. To understand the experiences of patients receiving HaH care and their caregivers; and
4. To understand the experiences of clinicians providing HaH in providing such care.

Further exploratory objectives include:

1. To identify factors that potentially influence the decisions of patients to accept HaH care, such as patient demographics, family and social setup, or perspectives of home-based care;
2. To describe the use of telehealth platforms for vital signs monitoring and teleconsultation that was used within the intervention arm; and
3. Study population

3.1 Setting

We study will recruit 147 patients in the intervention group and 147 patients in the control group from 2 sites: National University Hospital (NUH) and Alexandra Hospital (AH). Patients will be recruited from both AH and NUH with no restrictions of proportion from each center. There are no restrictions based on race of the subject. We will exclude children as this is an adult medical service.

3.2 Recruitment

3.2.1 Recruitment Process

Study personnel will screen through the electronic health record of all patients newly admitted overnight every working weekday in the following settings:

* NUH EMD Lodgers
* NUH Acute Medical Unit (AMU)
* NUH General Medicine Wards
* NUH Cardiology Wards
* AH wards under General Medicine (GM)

Patients thought to be suitable by the research assistant will be confirmed by the NUHS@Home consultant for clinical criteria, who will subsequently discuss with the primary physician regarding eligibility.

Patients who are subsequently enrolled into the NUHS@Home programme will be approached for consent to be in the hospital-at-home cohort. The NUHS@Home team will be activated. Patients will be sent home via ambulance, where they will be reviewed by a NUHS@Home nurse. Intravenous therapies, pillboxes for medication, remote monitoring software, and telecommunication tools will be set up as indicated. NUHS@Home doctors will visit at least once daily, and nurses at least twice daily as required. Therapists will conduct home visits as necessary. The NUHS@Home team is available 24/7. When conventional discharge criteria are met, the patient will be discharged. The NUHS@Home clinical team will be under clinical governance of Division of Advanced Internal Medicine at NUH and patients will be considered 'inpatients' throughout the treatment period.

Patients who are suitable for NUHS@Home programme but the programme has no bed capacity will be approached for consent to be in the control cohort. There will be no change to the patient's clinical management.

Patients who were offered but declined enrolments inot the NUHS@Home programme will be approached for consent to be in the rejected cohort. There will be no change to the patient's clinical management.

3.2.2 Consent

If the patient has capacity, the study team will go through the study information with the patient and caregiver (which will cover the process for recruitment and the randomisation process) and take written informed consent. If the patient requests, their main spokespersons will be involved in the discussion. If the patient has no capacity to consent, the main spokesperson will represent them in this scenario.

3.3 Inclusion and exclusion criteria are entered elsewhere in this protocol

3.4 Withdrawal Criteria

Patients may discontinue the intervention if they are transferred back to hospital during the treatment period.

3.5 Subject Replacement

Subjects who drop out will not be replaced.

4 Methods and Assessments

4.1 Study Visits

4.2.1 Screening Encounter

Patients which are potentially eligible would be screened both using the electronic health record and in person using a screening checklist to confirm eligibility.

4.2.2 Study Visits

Patients or their proxies who consent will undergo a baseline questionnaire. This includes baseline demographics, Barthel's score, assessment of health literacy, mini-COG, EQ-5D-5L and EQ-VAS. If a proxy is used, the same proxy will need to complete all subsequent questionnaires.

4.2.3 Final Study Visits

Patients will undergo a final questionnaire 14 days from enrolment. If a proxy was used for initial questionnaires, the same proxy will be used to complete the final questionnaire. This includes EQ-5D-5L, EQ-VAS, perception of care transitions and patient satisfaction survey. The visit will either be done in the clinic (if patients are coming for a clinic appointment) or over a phone call. Patients and caregivers in the intervention group will undergo an additional survey.

Patients in the 'rejected cohort' will not undergo this questionnaire.

4.2.4 Post Study Follow up and Procedures

30 days from discharge, the study team will collect patient outcomes from all 3 cohorts from the electronic medical record. Every 3 months, the study team will extract billing data for a list of itemised consumables and their associated cost to the patient. Patients will not be involved in this data collection.

5 Measurements

5.1 Primary and secondary outcomes are detailed elsewhere in this protocol

5.2 Baseline Characteristics

The following baseline characteristics will be measured at enrolment:

* Demographics (age, sex, ethnicity)
* Socioeconomic factors (occupation, income group, marital status, residence type, highest education level)
* Diagnosis at enrolment
* Number of hospitalisations in the last 12 months
* Home environment (who patients live with, main caregiver, housing type)
* Functional status (Barthel's Index , I-ADLs, assistance to doctor)
* NEWS score at enrolment
* Charlson Comorbidity Index at enrolment
* Clinical Frailty Score (at baseline) rated by NUHS@Home physician
* Cognitive impairment using Mini-COG
* Health Literacy using screening questions
* EQ-5D-5L

5.4 Process Evaluation

5.4.1 Process Measures

The following processes will also be measured in both groups from chart review:

* Number of appointments reduced upon discharge
* Number of referrals to community services
* Number of handovers to transitional care
* Number of patient and family education sessions done
* Number of unplanned physician encounters ("call-to-see-patient" or CTSPs), during and after office hours
* Number of days that patients received:

  * Vital signs monitoring
  * BSL monitoring
  * Wound dressing
  * Intravenous medication
  * Intravenous drip
  * Nebuliser therapy
  * Sliding scale insulin
  * Phlebotomy
* Whether patients received the following after enrolment:

  * Imaging
  * Endoscopy
  * Interventional radiology
  * Referral to medical speciality
  * Referral to non-medical specialty
* Discharged with written instructions or educational material
* Referral to advanced care planning
* Follow up in 72 hours from discharge

5.4.2 Disease specific quality indicators

Disease specific quality indicators will be measured for the common diagnoses that the investigators anticipate, and where established quality indicators exist.

* For heart failure :

  * ACEI/ARB or ARNI at discharge
  * Evidence Specific Beta blockers at discharge
  * Measurement or plan for measurement of LV function
  * Post-discharge appointment for heart failure
  * Adult smoking cessation advice
  * Influenza and pneumococcal vaccination
  * 30-day readmission for heart failure
* For COPD :

  * Initiation of long term oxygen therapy if appropriate
  * Identification for pulmonary rehabilitation
  * Antibiotics given
  * Glucocorticoids given
  * Appropriate prescription of relieving bronchodilators on discharge
  * Inhaler technique assessed
  * 30-day readmission for COPD exacerbation
* For urinary tract infection :

  * Urine culture performed
  * Prescribe empirical therapy according to hospital guidelines or previous cultures
  * Change to pathogen directed therapy with culture results are available
  * Change from intravenous to oral therapy in 48-72h on basis of clinical condition
  * Change catheter for long term in dwelling catheter
* For pneumonia :

  * Adult smoking cessation advice
  * Influenza and pneumococcal vaccination
  * Oxygen received if hypoxic
  * Conversion from intravenous to oral therapy when clinically improving, haemodynamically stable and tolerating orally

5.4.3 Intervention-specific Process Measures

The following processes will also be measured to examine fidelity of the programme:

* Response time for out-of-hour home visits
* Number of unexpected telephone calls & staff visits
* Number of medication reviews done with patient and family
* Number of patients transferred back to acute hospital
* Number of home visits by doctor and duration of each
* Number of home visits by nurse and duration of each
* Number of home visits by allied health and duration of each
* Number of home visits by caregivers and duration of each
* Number of virtual visits by doctor and duration of each
* Number of virtual visits by nurse and duration of each
* Number of virtual visits by allied health and duration of each

5.4.4 Stakeholder Perspectives Using a Qualitative Approach

Patients who are eligible and enrolled into the NUHS@Home Programme will be recruited for this study. They will also be asked if their family member/caregiver (excluding hired domestic help) might be interested to participate in the in-depth semi-structured interviews.

Study Design

The focused ethnography approach is adopted to elicit situated experiences of patients receiving care at home and the perceptions of caregivers and care providers in regard to facilitators and barriers to this new care model. Participant observations of care practices at home and interviews with the three parties including patients, caregivers and the staff will be undertaken. Analysis will be conducted using constant comparison technique to compare incidents applicable to each theme.

Observations will be carried out at participants' home by adopting 'observer as participant' role (Gold, 1958), where observations will be favored over participation. Interview guide will be adopted from the initial qualitative interviews and will focus on the following areas: Patients experiences of receiving the care at home: Caregivers and staff's perceptions of providing the care at home; Facilitators and barriers of receiving/providing care via HaH model and specific questions in regard to the rich points of social interaction observed in the field.

The following themes will be explored from the patient and their caregivers:

* Describe their experience of being admitted to the Hospital at Home programme.
* What, if any, are the benefits they have experienced during Hospital at Home?
* What, if any, are the disadvantages and drawbacks they have experienced during Hospital at Home?
* Did this program meet their expectations? Why or why not?
* Would they choose to be transferred to Home Hospital again if needed hospitalisation in the future? Why or why not?
* How did they feel about the vital signs monitoring setup at home?
* What, if any, is their experience of video or phone calls from the doctor during hospital at home?
* What, if any, is their experience with private doctors or nurses that attended to them during their stay?
* Any suggestions for the future development of Home Hospital?

Interviews will be audio-recorded and will last approximately 30-60 minutes. The interviews will focus on understanding the experiences of patients, caregivers and care providers on their perceptions of the HaH intervention program.

The total number of interviews required will depend on data saturation, estimated to involve 20-30 patients and 20-30 caregivers.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to one of the following wards:

   1. Episodic short stay patients

      * NUH Extended Diagnosis and Treatment Unit (EDTU)
      * AH Extended Diagnosis and Treatment Unit (EDTU)
      * NUH Acute Medical Unit (AMU)
   2. Long stay patients requiring ongoing treatment or monitoring

      * NUH general medicine wards
      * AH general medicine wards
   3. Speciality specific treatment and monitoring with a protocolised approach

      * Fluid overload admissions from NUH cardiology service
      * Fluid overload admissions from NUH nephrology service
2. ≥ 21 years old
3. Lives within the Western Cluster of Singapore (pre-specified list of postcodes)
4. Requires continued hospitalisation

   * The EDTU is a ward within the emergency department that patients can stay for up to 24hours for diagnosis and treatment and meant for discharge after. Some of these patients subsequently require hospital admission, which would be the target group for the pilot. The AMU is a short-stay ward at NUH which aims to discharge patients within 72 hours of stay.

Exclusion Criteria:

1. Lives in nursing home
2. Suitable for discharge to other community programmes
3. Planned for discharge the next day (D-1)
4. Haemodynamic instability defined as NEWScore >2 at time of recruitment (a NEWScore ≤2 in a local setting showed very low rates of transfer to intensive care and death in 24 hours )
5. Requires oxygen (long term oxygen therapy is acceptable)
6. Acute psychosis or suicidal intent
7. Need for negative pressure isolation
8. Anticipated to deteriorate
9. Planned for imaging, endoscopy, blood transfusion, cardiac stress test, surgery, interventional radiology procedures or ongoing non-medical specialist review
10. Need for intravenous controlled drugs (e.g. morphine)
11. Unable to establish venous access in emergency department
12. Current or former intravenous drug user
13. History of violence towards healthcare workers
14. Cannot provide meals at home
15. Does not have a bed, table and fridge at home
16. Patient or caregiver unable to use a phone
17. House is unsuitable for home visits and medical equipment
18. Unable to be homebound independent, or have a full-time caregiver to assist with daily activities if not homebound independent
19. Caregivers unable or unwilling to manage patient's care at home
20. Projected to require more than 2 weeks of rehab
21. For fluid overload cases, acute myocardial infarction within 5 days
22. Pregnant
23. Anticipated to require sliding scale insulin more than twice a day, where patient and/or caregiver are not able to measure BSL or administer insulin doses at home independently
24. Unable to understand simple instructions for oral self-administration of medication

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are enrolled into the NUHS@Home programme will be approached for consent to be in the hospital-at-home cohort.
  Patients who are suitable for NUHS@Home programme but the programme has no bed capacity will be approached for consent to be in the control cohort. There will be no change to the patient's clinical management.
  Patients who were offered but declined enrolments into the NUHS@Home programme will be approached for consent to be in the rejected cohort. There will be no change to the patient's clinical management.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Cost of care | At completion of intervention (an average of 7 days)
  The primary outcome is cost of care which the sum of the following:
  1. Itemised consumables
  2. Labour cost of physicians, estimated by the average time spent delivering care multiplied by standard salary (plus benefits) estimates of physicians' respective paygrades.
  3. Labour cost of nurses, estimated by the average time spent delivering care multiplied by standard salary (plus benefits) estimates of nurses' respective paygrades
  4. Labour cost of allied health (e.g. phlebotomists, physiotherapists) will be estimated by the average time spent delivering care multiplied by standard salary (plus benefits) estimates of their respective paygrades.
  5. Any additional costs incurred by the intervention group (e.g. telemonitoring, transport of blood tests) will be itemised as well.

SECONDARY OUTCOMES:
30-day readmission rate and attendance rate to emergency department | 30 days from completion of intervention (an average of 7 days)
  (planned and unplanned)
Death during treatment | At completion of intervention (an average of 7 days)
  (planned and unplanned)
30-day mortality | 30 days from enrolment
  (anticipated and unanticipated)
Iatrogenic events during treatment period | At completion of intervention (an average of 7 days)
  Composite outcome, total number of events including: falls, new delirium (not present at admission), DVT/PE, New pressure ulcer, Thrombophlebitis, Catheter associate UTI, New Clostridium Difficle Infection, New MRSA acquisition.
Number of bed days in hospital | At completion of intervention (an average of 7 days)
  Length of stay in hospital
Duration of treatment period | At completion of intervention (an average of 7 days)
  Length of stay
ICU/HD transfers | At completion of intervention (an average of 7 days)
  Escalation of care
Patient-reported activity during treatment period | At completion of intervention (an average of 7 days)
  Survey question
Improvement in HR-QoL (EQ-VAS) | Between enrolment and 14 days post-enrolment
  Change in EQ-VAS
Improvement in HR-QoL (EQ-5D) | Between enrolment and 14 days post-enrolment, a higher score means better outcome, ranging from 0 to 1
  Change in EQ-5D-5L index score
Quality-adjusted-life-days gained | Measurements from baseline, at completion of intervention (an average of 7 days) and 14 days post enrolment
  Measured by area-under-the-curve of EQ-5D-5L
Patient satisfaction score | At completion of intervention (an average of 7 days)
  National University Hospital inpatient satisfaction survey which is adapted from the Care Quality Commission (CQC), Picker Institute and National Research Corporation (NRC) Inpatient Core Questionnaire
Caregiver Burden (if applicable) | At completion of intervention (an average of 7 days)
  Short version Zarit Burden Inventory (ZBI)
Care transitions experience | Within a month after completion of intervention (an average of 7 days)
  Care Transitions Measure CTM-3

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Q Ko, MBBS MPH, Principal Investigator — National University Health Systems
Locations (2):
- Singapore (2):
  - Alexandra Hospital, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goncalves-Bradley DC, Iliffe S, Doll HA, Broad J, Gladman J, Langhorne P, Richards SH, Shepperd S. Early discharge hospital at home. Cochrane Database Syst Rev. 2017 Jun 26;6(6):CD000356. doi: 10.1002/14651858.CD000356.pub4. PMID 28651296
- [Background] Caplan GA, Sulaiman NS, Mangin DA, Aimonino Ricauda N, Wilson AD, Barclay L. A meta-analysis of "hospital in the home". Med J Aust. 2012 Nov 5;197(9):512-9. doi: 10.5694/mja12.10480. PMID 23121588
- [Background] Shepperd S, Iliffe S, Doll HA, Clarke MJ, Kalra L, Wilson AD, Goncalves-Bradley DC. Admission avoidance hospital at home. Cochrane Database Syst Rev. 2016 Sep 1;9(9):CD007491. doi: 10.1002/14651858.CD007491.pub2. PMID 27583824
- [Background] Qaddoura A, Yazdan-Ashoori P, Kabali C, Thabane L, Haynes RB, Connolly SJ, Van Spall HG. Efficacy of Hospital at Home in Patients with Heart Failure: A Systematic Review and Meta-Analysis. PLoS One. 2015 Jun 8;10(6):e0129282. doi: 10.1371/journal.pone.0129282. eCollection 2015. PMID 26052944
- [Background] Jeppesen E, Brurberg KG, Vist GE, Wedzicha JA, Wright JJ, Greenstone M, Walters JA. Hospital at home for acute exacerbations of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 May 16;2012(5):CD003573. doi: 10.1002/14651858.CD003573.pub2. PMID 22592692
- [Background] Federman AD, Soones T, DeCherrie LV, Leff B, Siu AL. Association of a Bundled Hospital-at-Home and 30-Day Postacute Transitional Care Program With Clinical Outcomes and Patient Experiences. JAMA Intern Med. 2018 Aug 1;178(8):1033-1040. doi: 10.1001/jamainternmed.2018.2562. PMID 29946693
- [Background] Echevarria C, Gray J, Hartley T, Steer J, Miller J, Simpson AJ, Gibson GJ, Bourke SC. Home treatment of COPD exacerbation selected by DECAF score: a non-inferiority, randomised controlled trial and economic evaluation. Thorax. 2018 Aug;73(8):713-722. doi: 10.1136/thoraxjnl-2017-211197. Epub 2018 Apr 21. PMID 29680821
- [Background] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232
- [Background] Montalto M. The 500-bed hospital that isn't there: the Victorian Department of Health review of the Hospital in the Home program. Med J Aust. 2010 Nov 15;193(10):598-601. doi: 10.5694/j.1326-5377.2010.tb04070.x. PMID 21077817
- [Derived] Ko SQ, Rahman N, Chai JH, Goh J, Luo N, Shi L, Lai YF, Soong JTY, Chan DKW, Peh ALT, Kuan WS, Lim YW. Hospital-at-home versus hospital admission for acute care in Singapore: a prospective quasi-experimental study on cost, utilisation and clinical outcomes. BMC Health Serv Res. 2026 Jan 20. doi: 10.1186/s12913-025-13938-5. Online ahead of print. PMID 41559634